CLINICAL TRIAL: NCT00925691
Title: Comparison of SEPTal and Apical Pacing Sites in PerManent Right Ventricular Pacing
Acronym: SEPTAL-PM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCB : 2008-A01027-48; LOC / 05-12 (Other: Rennes University Hospital)
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Atrioventricular Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- APICAL (Active Comparator): implantation at the apex
  Interventions: Device: RV lead
- SEPTAL (Experimental): implantation at the interventricular septum
  Interventions: Device: RV lead

INTERVENTIONS:
Device: RV lead — The RV lead is implanted at the apex or at the interventricular septum

SUMMARY:
The SEPTAL-PM study is aimed to compare the right ventricular apical and right ventricular septal position of the right ventricular lead in patients implanted with a pacemaker for conventional anti-bradycardia pacing indications requiring permanent right ventricular pacing ; the primary endpoint is the evolution of the left ventricular ejection fraction assessed by contrast echocardiography at 18-months follow-up.

DETAILED DESCRIPTION:
Classically the right ventricular pacing (RV) lead position is the RV apex. Several small studies suggested that the septal position which provided a more physiological conduction pattern would improve left ventricular function and dimensions and the patients' outcome.

The SEPTAL-PM study is a parallel randomized prospective simple-blinded and multicenter national study with a follow-up duration of 18 month. A total of 180 patients will be enrolled.

It was designed to demonstrate that in patients requiring permanent RV pacing for high degree atrio-ventricular conduction disorders the septal pacing would preserve the LVEF and LV dimensions but also the quality of life and the exercise tolerance.

The primary endpoint is the evolution of the LVEF assessed by contrast echocardiography. The secondary endpoints are: the quality of life SF 36 questionnaire, the NYHA class, the 6-minute-walk test, the QRS duration, the LV end-systolic and diastolic volumes, the NT-pro BNP, MMP 2-9 and TIMP-1 dosages, stimulation and detection ventricular thresholds.

Other reported parameters are: the probes position and electric parameters, all causes of mortality, cardiovascular mortality, hospitalisations for cardiovascular causes, serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Written informed consent.
* Permanent cardiac pacing indication for high degree AV block with ventricular rate less than 50 bpm according to the current guidelines of the European Society of Cardiology .
* Patients with sinus rhythm or permanent atrial fibrillation.

Non-inclusion Criteria:

* Indication for cardiac resynchronization.
* Indication for Intra cardiac defibrillators (ICD).
* Indication for AV node ablation for patients with atrial fibrillation.
* Patients already implanted with a pacemaker or an ICD.
* Myocardial infarction within the previous month.
* Surgically treated valvulopathy.
* Tricuspid Valve prothesis
* Cardiac surgery or coronary revascularization planned or within the 3 last months.
* Life expectancy less than 18 months.
* Pregnancy.
* Disability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 18 months

SECONDARY OUTCOMES:
Quality of life questionnaire SF 36 | 18 months
NYHA class | 1, 6, 12, 18 months
6-minute-walk test | 1, 18 months
LV end-systolic and diastolic volumes | 18 months
QRS duration, | 1, 6, 12, 18 months
Evolution of cardiac remodeling markers: MMP2-9 and TIMP-1 and NT-pro BNP dosage | 18 months
All causes and cardiovascular mortality, hospitalizations for cardiovascular cause | 18 months
Serious adverse events | 18 months
Stimulation and detection ventricular thresholds | 1, 6, 12, 18 months
Probes position and electric parameters | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Leclercq, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - CHU d'Angers, Angers
  - Service de cardiologie-CHU de Brest, Brest
  - Service de cardiologie-CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes

REFERENCES:
- [Result] Galand V, Martins RP, Donal E, Behar N, Crocq C, Soulie GG, Degand B, Garcia R, Solnon A, Lande G, Probst V, Marjaneh F, Mansourati J, Dupuis JM, Laviolle B, Leclercq C. Septal versus apical pacing sites in permanent right ventricular pacing: The multicentre prospective SEPTAL-PM study. Arch Cardiovasc Dis. 2022 May;115(5):288-294. doi: 10.1016/j.acvd.2021.12.007. Epub 2022 Feb 19. PMID 35221255